CLINICAL TRIAL: NCT01562249
Title: Rehabilitative Management of Mastication After Orthognathic Surgery: A Randomized Controlled Trial
Brief Title: Rehabilitative Management of Mastication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ORTHOGSURG01
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Surgery; Malocclusion
Keywords: clinical evaluation; controlled clinical trial; electromyography; exercise program; motor control
MeSH Terms: conditions — Malocclusion | interventions — Counseling; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental group (Experimental): Inclusion criteria were: Skeletal Class III orthognathic surgery patients; adults (age above 18 years), agreement to perform orthognathic surgery and to undergo all of the necessary procedures determined by the multidisciplinary team (i.e. orthodontic preparation, clinical orofacial myofunctional and electromyographic assessment, surgery, post surgery orthodontic treatment, post surgery clinical orofacial myofunctional and electromyographic assessment and orofacial myofunctional treatment when necessary). Exclusion criteria were: previous orthognathic surgery; previous head and neck surgery; neurologic and/or systemic diseases; facial trauma; syndromes; cognitive impairment; and communication and hearing deficits.
  Interventions: Other: orofacial myofunctional treatment protocol
- Instruction Group (Active Comparator): Inclusion criteria were: Skeletal Class III orthognathic surgery patients, adults (age above 18 years), agreement to perform orthognathic surgery and to undergo all of the necessary procedures determined by the multidisciplinary team (i.e. orthodontic preparation, clinical orofacial myofunctional and electromyographic assessment, surgery, post surgery orthodontic treatment, post surgery clinical orofacial myofunctional and electromyographic assessment and orofacial myofunctional treatment when necessary). Exclusion criteria were: previous orthognathic surgery; previous head and neck surgery; neurologic and/or systemic diseases; facial trauma; syndromes; cognitive impairment; and communication and hearing deficits.
  Interventions: Other: counseling
- Control group (No Intervention): Inclusion criteria for this group were: adults (age above 18 years); absence of stomatognathic system alterations; absence of alterations in the scapular region; complete permanent dentition (absence/extraction of the third molar was accepted); Skeletal and Angle's Class I facial pattern; and absence of malocclusion. Exclusion criteria were: previous orthodontic treatment; and history of previous oral motor intervention.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: orofacial myofunctional treatment protocol — Once a week for six weeks, the experimental group received a forty minutes session of orofacial myofunctional treatment. A home exercise program was prescribed during each session. The protocol implies in continuous and daily practices - participants were asked to perform exercises at least three times a day. After the first six weeks, the experimental group underwent four sessions for maintenance purposes (two sessions twice a month and two sessions once a month). The total treatment duration was of five months.
  Other Names: rehabilitative orofacial myofunctional protocol
  Arms: Experimental group
Other: counseling — The instruction group underwent two supervised forty minutes therapy sessions along the six weeks following surgery. These sessions involved the perception of the stomatognathic system, especially in terms of adequate performance during mastication. Specific exercises were not given and patients were instructed to try to reproduce the adequate pattern of mastication at all meals (i.e. alternated bilateral, with lip closure; with coordination activity of the tongue and mandible).
  Other Names: supervised instruction
  Arms: Instruction Group
Other: Control Group — As the sEMG test-retest is a critical issue, participants of CG were also tested in two distinct moments (testing occurred with 1 year interval) in order to verify possible changes in the sEMG measurements as a result of retesting.
  Other Names: healthy individuals; no intervention
  Arms: Control group

SUMMARY:
The purpose of this study is to verify the effectiveness of a systematic rehabilitative program for mastication in patients submitted to orthognathic surgery.

DETAILED DESCRIPTION:
Orthognathic surgery can produce complications during the postoperative period - i.e. situations of acute pain and inflammation - as a consequence of fractures and incisions in the mucosa. The inadequate management of soft tissue and prolonged surgical time could be the causes of acute facial oedema, hematoma and ecchymosis in the face and neck, as well as functional disorders involving swallowing and breathing, which can affect patients' integrity.

Despite the fact that decreased muscular extensibility and strength, increased muscular fatigability, hipomobility, and alteration of the biomechanical efficiency and length of the masticatory muscles are documented clinical consequences, no systematic method of obviating such problems through muscular rehabilitation has yet been published

ELIGIBILITY:
Inclusion Criteria:

* Skeletal Class III orthognathic surgery patients
* adults (age above 18 years)
* agreement to perform orthognathic surgery
* agreement to undergo all of the necessary procedures determined by the multidisciplinary team

Exclusion Criteria:

* previous orthognathic surgery
* previous head and neck surgery
* neurologic and/or systemic diseases
* facial trauma
* syndromes
* cognitive impairment
* communication and hearing deficits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evidence of clinical improvement in mastication after oral-motor rehabilitative program | within the first year after surgery (plus or minus 2 weeks)
  improvement is verified through a clinical orofacial myofunctional evaluation using a standardized protocol with scores (orofacial mobility, masticatory/deglutition clinical performance, jaw movements) and by variations in the activation of the masseter and temporal muscles (surface electromyography)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia RF Andrade, Professor, Study Chair — School of Medicine, University of São Paulo; Laura D Mangilli, Ph.D., Principal Investigator — School of Medicine, University of São Paulo
Locations (1):
- Hospital das Clinicas, University of São Paulo, São Paulo, São Paulo, Brazil